CLINICAL TRIAL: NCT05183789
Title: Serum Levels of Interleukins 6 and 8 in Malnourished Children With Acute Diarrhea
Brief Title: IL6&8 in Malnourished Children With Acute Diarrhea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Motaz Mohamed Hassan, Pediatric Resident, Sohag University
Other Study IDs: IL6&8
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Acute Diarrhea; Severe Acute Malnutrition; Acute Gastroenteritis
Keywords: Children; Acute diarrhea; Severe acute malnutrition; Interleukins; Cytokines
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Malnourished children with acute diarrhea
  Interventions: Diagnostic Test: Evaluation of serum levels of IL-6 and IL-8
- Control: Non-malnourished children with acute diarrhea
  Interventions: Diagnostic Test: Evaluation of serum levels of IL-6 and IL-8

INTERVENTIONS:
Diagnostic Test: Evaluation of serum levels of IL-6 and IL-8 — Evaluation of serum levels of IL-6 and IL-8 by Luminex Assay (multiplexed ELISA kits).

SUMMARY:
Cytokines, such as IL-6 and IL-8 can be used as markers of acute infections, including acute gastroenteritis. However, there have been no previous studies on the levels of IL-6 and IL-8 in malnourished children with acute diarrhea. This study aims to evaluate serum levels of interleukins 6 and 8 in malnourished children with acute diarrhea.

DETAILED DESCRIPTION:
Acute gastroenteritis remains a common health problem among children worldwide with significant morbidity, mortality, and economic burden. Diarrheal diseases account for more than half-million deaths of children under 5 years old every year, most of which take place in low- and middle-income countries (LMICs). Moreover, diarrheal diseases are a leading cause of emergency visits and hospitalization. According to the WHO, acute diarrhea is classified into acute watery diarrhea, acute bloody diarrhea (dysentery), persistent diarrhea, and diarrhea with severe malnutrition. Acute watery diarrhea is the most common category in both high and LMICs. Viral infections (e.g., rotavirus, norovirus, adenovirus) are the leading causes of acute watery diarrhea in children (up to 90% of cases), while bacteria (e.g., shigella, salmonella, Campylobacter, enterotoxigenic E. coli) and parasites (e.g., Cryptosporidium, Giardia, and E. histolytica) account for the remainder of cases.

Cytokines can be used as markers of acute infections, including acute gastroenteritis. Interleukin-6 (IL-6) is produced by lymphoid and non-lymphoid cells and plays important role in regulation of immunity, acute-phase response, and hematopoiesis; IL-6 has a well-known role in the defense mechanism in acute gastroenteritis. Interleukin-8 (IL-8) functions in chemotaxis of inflammatory cells, such as neutrophils and lymphocytes, to the site of inflammation, Both IL-6 and IL-8 are critical for immunity against mucosal infections; they are released from the epithelial cells of the gastrointestinal tract to mount its inflammatory responses to infectious agents at local and systemic levels.

Some studies investigated the role of IL-6 and IL-8 as biomarkers for acute diarrhea in children. Results showed significantly increased serum levels of IL-6 and IL-8 in children with acute GE compared with healthy controls. Moreover, IL-6 is significantly elevated in bacterial gastroenteritis in comparison to viral gastroenteritis. However, none of these studies included children with severe acute malnutrition.

Severe acute malnutrition (SAM) is a severe form of malnutrition resulting from inadequate or poor quality dietary intake. This is a serious public health problem, particularly in developing countries. SAM can be classified into marasmus, characterized by overt loss of subcutaneous fat and muscle mass, and Kwashiorkor, characterized by bilateral pitting edema of lower limbs.

Malnutrition is one of the most common causes of impaired immune function in children. Malnutrition leads to defects of phagocytosis, chemotactic function of neutrophils and monocytes, complement system and opsonization, and the function of antigen presenting cells.

As part of its negative impact on immune system, SAM may impair acute phase inflammatory response, including cytokines. In vitro studies showed that peripheral blood mononuclear cells from malnourished children have reduced ability to produce cytokines, such as IL-1, IL-6, IL-8, and tumor necrosis factor alpha. Some studies showed that children with SAM have significantly lower levels of IL-6 and IL-8 compared with healthy controls [8]. In contrast, other studies showed similar or higher levels of pro-inflammatory cytokines in malnourished children compared with healthy controls.

To the best of our knowledge, there have been no previous studies on the levels of IL-6 and IL-8 in children with SAM and acute diarrhea.

The aim of this study is to evaluate serum levels of interleukins 6 and 8 in malnourished children with acute diarrhea.

ELIGIBILITY:
Group 1: Cases (Malnourished children with acute diarrhea)

Inclusion Criteria:

* Age: 6 months to 5 years.
* Severe acute malnutrition. Infants and children who are 6-59 months of age and have a mid-upper arm circumference < 115 mm or a weight for height/length <-3 Z-score of the WHO growth standards or have bilateral edema.
* Acute diarrhea: Defined according to WHO criteria as the "passage of loose or watery stools at least three times in a 24 h period", lasts less than 14 days, with or without fever or vomiting, but considering the importance of change in stool consistency rather than frequency, and the usefulness of parental insight in deciding whether children have diarrhea or not.

Exclusion Criteria:

* History of antibiotic therapy in the last 72 hours.
* Acute diarrhea in association with systemic infections
* Malignancy
* Chronic diarrhea
* Autoimmune and autoinflammatory diseases.
* Chronic renal/liver failure
* Diabetes mellitus

Group 2: Control (Non-malnourished children with acute diarrhea)

Inclusion Criteria:

* Healthy children aged 6 months to 5 years.
* Acute diarrhea

Exclusion Criteria:

* Malnutrition or obesity
* History of antibiotic therapy in the last 72 hours.
* Acute diarrhea in association with systemic infections
* Malignancy
* Chronic diarrhea
* Autoimmune and autoinflammatory diseases.
* Chronic renal/liver failure
* Diabetes mellitus

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children presented to the Pediatric Department and Outpatient Clinic at Sohag University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Serum level of Interleukin 6 | Within the first 3 days of acute diarrhea
  Difference in serum level of interleukin 6 between cases and control groups
Serum level of Interleukin 8 | Within the first 3 days of acute diarrhea
  Difference in serum level of interleukin 8 between cases and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim A Sadek, MD, PhD, Study Chair — Faculty of Medicine, Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Immediately after publication
Access Criteria: Researchers working on relevant field

REFERENCES:
- [Background] Zaki MES, Alsayed MAL, Shrief R. Study of the diagnostic value of interleukin-6 and interleukin-8 in children with acute gastroenteritis. Germs. 2020 Mar 2;10(1):27-33. doi: 10.18683/germs.2020.1182. eCollection 2020 Mar. PMID 32274357
- [Background] Rankin JA. Biological mediators of acute inflammation. AACN Clin Issues. 2004 Jan-Mar;15(1):3-17. doi: 10.1097/00044067-200401000-00002. PMID 14767362
- [Background] Svanborg C, Godaly G, Hedlund M. Cytokine responses during mucosal infections: role in disease pathogenesis and host defence. Curr Opin Microbiol. 1999 Feb;2(1):99-105. doi: 10.1016/s1369-5274(99)80017-4. PMID 10047563
- [Background] Chen SM, Lin CP, Tsai JD, Chao YH, Sheu JN. The significance of serum and fecal levels of interleukin-6 and interleukin-8 in hospitalized children with acute rotavirus and norovirus gastroenteritis. Pediatr Neonatol. 2014 Apr;55(2):120-6. doi: 10.1016/j.pedneo.2013.05.008. Epub 2013 Jul 27. PMID 23899552
- [Background] Ibrahim MK, Zambruni M, Melby CL, Melby PC. Impact of Childhood Malnutrition on Host Defense and Infection. Clin Microbiol Rev. 2017 Oct;30(4):919-971. doi: 10.1128/CMR.00119-16. PMID 28768707
- [Background] Marginean CO, Man L, Pitea AM, Man A, Marginean CL, Cotoi OS. The assessment between IL-6 and IL-8 and anthropometric status in malnourished children. Rom J Morphol Embryol. 2013;54(4):935-8. PMID 24398988
- [Background] Dulger H, Arik M, Sekeroglu MR, Tarakcioglu M, Noyan T, Cesur Y, Balahoroglu R. Pro-inflammatory cytokines in Turkish children with protein-energy malnutrition. Mediators Inflamm. 2002 Dec;11(6):363-5. doi: 10.1080/0962935021000051566. PMID 12581501
- [Background] Malave I, Vethencourt MA, Pirela M, Cordero R. Serum levels of thyroxine-binding prealbumin, C-reactive protein and interleukin-6 in protein-energy undernourished children and normal controls without or with associated clinical infections. J Trop Pediatr. 1998 Oct;44(5):256-62. doi: 10.1093/tropej/44.5.256. PMID 9819485